CLINICAL TRIAL: NCT04808635
Title: The Predictors of Depression and Burnout Among Surgical Residents: A Cross-sectional Study From Kuwait
Status: Completed | Type: Observational
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Waleed burhamah, Dr. Waleed burhamah, General surgery resident MKH, Ministry of Health, Kuwait
Other Study IDs: MOHKWMKH21
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- general surgery residents
  Interventions: Other: no intervention, this is a cross sectional questionnaire based study.
- orthopedic surgery residents
  Interventions: Other: no intervention, this is a cross sectional questionnaire based study.
- urology residents
  Interventions: Other: no intervention, this is a cross sectional questionnaire based study.
- OBGYN residents
  Interventions: Other: no intervention, this is a cross sectional questionnaire based study.

INTERVENTIONS:
Other: no intervention, this is a cross sectional questionnaire based study. — no intervention, this is an observational cross sectional study

SUMMARY:
To assess the prevalence and risk factors for depression and burnout among residents across surgical specialties in Kuwait.

DETAILED DESCRIPTION:
This is a questionnaire based cross-sectional study conducted in Kuwait from jan 2021- February 2021 An online questionnaire was sent to the residents enrolled to the surgical residency programs in Kuwait. Residency training in Kuwait provides programs in both medical and surgical specialties. Specialties included in our cohort were: general surgery, orthopedic surgery, urology, neurosurgery, Obstetrics and Gynecology and otolaryngology.

The email sent to our participants included an invitation letter detailing the reason behind the questionnaire and that it is confidential and anonymous. Consent was obtained from participants.

Variables:

Variables collected included; age, gender, marital status, smoking history, exercise, specialty, year of training, on-call frequency, assessment of burnout and assessment of depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

- residents enrolled in surgical training in Kuwait. Across all surgical specialties From R1-R5

Exclusion Criteria:

Recently accepted candidates that have not yet started residency.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: surgical residents across 4 specialties.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Symptoms of depression were assessed using the 9-item Patient Health Questionnaire (PHQ-9) score | 1 month
  (PHQ-9) score, a self-report questionnaire that is commonly used as a screening tool for depression. It is composed of 9 questions assessing the frequency of depressive symptoms on a 4-point Liker-scale ranging from 0 (never) to 3 (nearly every day). The total score was calculated for each patient and was interpreted as follows: minimal (1-4), mild (5-9), moderate (10-14), moderately severe (15-21), severe (20-27). A standard cutoff of score of 10 was used, indicating a diagnosis of depression.
Burnout symptoms were assessed using 9-item form of the Maslach Burnout Inventory - Human Services Survey (aMBI-HSS) | 1 month
  The aMBI is a 9-item questionnaire each question is rated on a 7-point Liker scale ranging from 0 to 6, which indicates the frequency of symptoms in question. Response options include; Every day, A few times a week, Once a week, A few times a month, Once a month, A few times a year, or Never. The questions grouped into 3 subscales (emotional exhaustion EE, depersonalization D and personal accomplishment PA) are evaluated and scored separately with each score ranging from 0 to 18. We used the cut off points set by Lebares et al. for EE and D. The cut off points for high burnout among U.S. surgery residents were: EE score ≥ 9 and D score ≥ 6. A PA score ≤ 12 was chosen as a cut-off for high burnout.

CONTACTS AND LOCATIONS:
Locations (1):
- Mubarak al Kabeer hospital, Kuwait City, Outside U.S./Canada, Kuwait

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code